CLINICAL TRIAL: NCT05131984
Title: Ocrelizumab Treatment Access and Outcomes by Gender, Race, and Socio-economic Status in Multiple Sclerosis Patients: Real World Investigation
Brief Title: Ocrelizumab Access by Socio-Economic Status
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genentech, Inc. (Industry); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Maria Houtchens, Neurologist, Director of the Clinical Care, Multiple Sclerosis Center, Brigham and Women's Hospital
Other Study IDs: 2021P002772
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Multiple Sclerosis patients on Ocrelizumab at Brigham and Women's Hospital: All MS patients at the Brigham MS Center who have been diagnosed with relapsing remitting multiple sclerosis (RRMS) or primary progressive multiple sclerosis (PPMS), ages 18 or older, on Ocrelizumab for at least one year and have received at least 3 treatments (two loading treatments of 300mg each, and one full dose treatment of 600 mg), who have been followed at these institutions for clinical care and brain and/or spinal cord MRI, and who have received Ocrelizumab infusions at these institutions for the duration of the study period.
  Interventions: Drug: Ocrelizumab
- Multiple Sclerosis patients on Ocrelizumab at Boston Medical Center: All MS patients at the Boston Medical Center MS Clinic who have been diagnosed with RRMS or PPMS, ages 18 or older, on Ocrelizumab for at least one year and have received at least 3 treatments (two loading treatments of 300mg each, and one full dose treatment of 600 mg), who have been followed at these institutions for clinical care and brain and/or spinal cord MRI, and who have received Ocrelizumab infusions at these institutions for the duration of the study period.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — At least 3 treatments (two loading treatments of 300mg each, and one full dose treatment of 600 mg over the course of 1 year

SUMMARY:
The primary aim of this project is to determine whether there are differences in access to, efficacy and tolerability of Ocrelizumab in men and women of different racial and ethnic origins and socio-economic backgrounds with RRMS and PPMS in two large academic MS Centers with a high volume of patients on Ocrelizumab. The study is a retrospective analysis of multiple sclerosis patients cared for at Brigham and Women's Hospital and Boston Medical Center who were treated with Ocrelizumab during the 4 year study period.

DETAILED DESCRIPTION:
This study will be a two-center retrospective/observational analysis with data collected from the Research Patient Data Registry (RPDR), Brigham Multiple Sclerosis Center Patient Database (Oracle), and Boston Medical Center MS Clinic Database (BMC-MS).

Using the Oracle database, BMC-MS database and electronic medical records (EPIC), the investigators will capture all MS patients who satisfy inclusion criteria. This study will collect age, sex, race, socio-economic status by residence zip code, disease duration, previous treatment, current treatment status, the reason for discontinuing or switching to another treatment, expanded disability status scale (EDSS), and functional systems scores (FSS) where available.

Additionally, the investigators will collect the date, dose, and interval between each ocrelizumab infusion, as well as any pertinent laboratory values and MRI scan results.

ELIGIBILITY:
Inclusion Criteria:

* All MS patients at the Brigham MS Center and Boston Medical Center MS Clinic who have been diagnosed with RRMS or PPMS, ages 18 or older, on Ocrelizumab for at least one year and have received at least 3 treatments (two loading treatments of 300mg each, and one full dose treatment of 600 mg), who have been followed at these institutions for clinical care and brain and/or spinal cord MRI, and who have received Ocrelizumab infusions at these institutions for the duration of the study period.

Exclusion Criteria:

* Simultaneous use of high dose monthly IV steroids,
* Secondary progressive MS (SPMS) disease category,
* Additional serious medical or neurologic co-morbid diseases,
* Additional concomitant immunosuppressive therapy of any kind,
* Additional concomitant MS-specific therapy (DMT) of any kind,
* Change of infusion or care site and absence of neurologic or imaging follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing remitting or primary progressive MS evaluated at Brigham and Women's Multiple Sclerosis Clinic or Boston Medical College Multiple Sclerosis Clinic between 03/2017 and 07/2021 who were started on ocrelizumab in that time period.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Time to treatment initiation | 03/2017 - 07/2021
  Time from diagnosis to Ocrelizumab treatment initiation in men and women of different racial and ethnic origins and socio-economic backgrounds with RRMS and PPMS.

SECONDARY OUTCOMES:
Annualized relapse rate | 12-24 months from ocrelizumab initiation
  Annualized relapse rate over 12 and 24 months in men and women of different racial and ethnic origins and socio-economic backgrounds in patients with RRMS.
MRI Changes | 12-24 months from ocrelizumab initiation
  New T2 and new T1 gadolinium enhancing lesions over 12 and 24 months in men and women of different racial and ethnic origins and socio-economic backgrounds in patients with RRMS.

OTHER OUTCOMES:
Adverse Effects | 03/2017 - 07/2021
  Evaluation of the prevalence of adverse effects in men and women of different racial and ethnic origins and socio-economic backgrounds with RRMS and PPMS.
Treatment Discontinuation | 03/2017 - 07/2021
  Evaluation of the reasons for and timing of discontinuation of treatment with ocrelizumab in men and women of different racial and ethnic origins and socio-economic backgrounds with RRMS and PPMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No